CLINICAL TRIAL: NCT04925193
Title: Personalized Selinexor-based Therapy for Relapsed/Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-2202.cc; P30CA046934 (NIH)
Record Dates: First submitted 2021-05-19; First posted 2021-06-14 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma in Relapse
MeSH Terms: interventions — selinexor; pomalidomide; daratumumab; carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 SPd (Experimental): * Selinexor 60 mg PO days 1, 8, 15
  * Pomalidomide 4 mg PO on days 1-21
  * Dexamethasone 40 mg PO or IV on days 1, 8, 15, 22
  * 28 day treatment cycles
  Interventions: Drug: Selinexor; Drug: Pomalidomide; Drug: Dexamethasone
- Arm 2 SDd (Experimental): * Selinexor 80 mg PO days 1, 8, 15
  * Daratumumab 1,800mg/30,000 units subcutaneous injection on days 1, 8, 15, 22 of cycles 1 and 2, days 1, 15 of cycles 3-6, day 1 of cycles >6
  * Dexamethasone 40 mg PO or IV days 1, 8, 15, 22
  * 28 day treatment cycle
  Interventions: Drug: Selinexor; Drug: Daratumumab; Drug: Dexamethasone
- Arm 3 SKd (Experimental): * Selinexor 80 mg PO days 1, 8, 15
  * Carfilzomib IV infusion 20 mg/m2 cycle 1, day 1, 56 mg/m2 cycle 1 day 8, 15. Cycle 2+ days 1, 8, 15.
  * Dexamethasone 40 mg IV or PO days 1, 8, 15, 22
  * 28 day treatment cycle
  Interventions: Drug: Selinexor; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Selinexor is an oral, first-in-class, slowly reversible, potent selective inhibitor of nuclear export (SINE) compound that specifically blocks exportin 1 (XPO1).
Drug: Pomalidomide — Oral Table
  Arms: Arm 1 SPd
Drug: Daratumumab — Injection
  Arms: Arm 2 SDd
Drug: Carfilzomib — Injection
  Arms: Arm 3 SKd
Drug: Dexamethasone — Oral tablet or injection

SUMMARY:
Selinexor (KPT-330, Xpovio) is a first in class selective inhibitor of nuclear export which has been approved for use in relapsed and refractory multiple myeloma (RRMM). This trial will seek to evaluate the outcomes achieved with selinexor based combination in RRMM selected by physician's choice and compared prospectively to ex vivo drug sensitivity testing results. Participants will be enrolled and assigned into one of the following treatment arms:

Arm 1: Selinexor + pomalidomide + dexamethasone (SPd)

Arm 2: Selinexor + daratumumab + dexamethasone (SDd)

Arm 3: Selinexor + carfilzomib + dexamethasone (SKd)

DETAILED DESCRIPTION:
This study is a single institution, open-label phase II study to evaluate the overall response rate achieved with selinexor and dexamethasone based three drug combination therapy, selected by physician's choice, in patients with relapsed/refractory multiple myeloma.

Patients with RRMM will be eligible for enrollment. During screening, in addition to standard of care disease assessments, participant's bone marrow aspirate will be evaluated using a novel ex vivo Myeloma Drug Sensitivity Testing platform (My-DST). The following agents will be eligible for physician's choice, and in parallel evaluated for sample sensitivity in MyDST: pomalidomide, carfilzomib and daratumumab. Agents will be tested individually, in combination with selinexor and in combination with selinexor and dexamethasone. Results from MyDST will be not be available to investigators at time of treatment assignment, but will be evaluated to better characterize test performance and relationship with treatment outcomes.

Investigators will assign patients to one of the following treatment combinations: Selinexor/Pomalidomide/Dexamethsone (SPd), Selinexor/Daratumumab/Dexamethasone (SDd) or Selinexor/Carfilzomib/Dexamethasone (SKd). Investigators will use patient specific considerations such as prior therapeutic exposures, response to / tolerance of prior therapies and comorbid conditions which may increase risk for toxicity with specific agents to guide expert judgement in selecting partner agent for selinexor and dexamethasone. Treatment will continue until progression of disease, unacceptable toxicity or death.

This study will evaluate if physician's choice partner drug selection for selinexor based combination therapy in RRMM will lead to an overall response rate of 75% or higher.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Willing and able to provide written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
4. Histologically confirmed diagnosis, measurable disease and evidence of disease progression of MM after 1 or more prior lines of therapy with either of:

   1. Documented evidence of PD after achieving at least SD for ≥ 1 cycle during a previous MM regimen (i.e., relapsed MM)
   2. ≤ 25% response (i.e, patient never achieved ≥ MR) or PD during or within 60 days from end of the most recent MM regimen (i.e., refractory MM)
5. Patients must have measurable disease as defined by at least one of the following:

   a) Serum M-protein ≥ 0.5 g/dL by serum protein electrophoresis (SPEP) or, for IgA myeloma, by quantitative IgA c) Urinary M-protein excretion at least 200 mg/24 hours d) Serum FLC ≥ 10 mg/dL, provided that FLC ratio is abnormal e) If no measurable disease by serum or urine, then the presence of a plasmacytoma of ≥ 2cm in one dimension prior to start of study can be used to follow response via radiologic imaging
6. Adequate hepatic function:

   f) Total bilirubin <1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of <3 × ULN), and g) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 × ULN.
7. Adequate renal function as determined by serum creatinine of ≤ 2 mg/dL OR estimated creatinine clearance of ≥ 20 mL/min, calculated using the Cockcroft and Gault formula (140 - Age) • Mass (kg)/ (72 • creatinine mg/dL); multiply by 0.85 if female.
8. Adequate hematopoietic function within 28 days prior to C1D1: absolute neutrophil count ≥1000/mm3, hemoglobin ≥8 g/dL and platelet count ≥100,000/mm3 (patients for whom <50% of bone marrow nucleated cells are plasma cells) or ≥50,000/mm3 (patients for whom ≥50% of bone marrow nucleated cells are plasma cells).

   1. Patients may receive hematopoietic growth factor support, including erythropoietin, darbepoetin, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), and platelet stimulators (eg, eltrombopag, romiplostim, or interleukin-11) at any time
   2. Patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study.
9. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 3 months following the last dose of protocol required therapies.

Exclusion Criteria:

1. Has received selinexor or another XPO1 inhibitor in a previous line of therapy
2. Has any concurrent medical condition or disease (eg, uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.) that is likely to interfere with study procedures.
3. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to Cycle 1 Day 1 (C1D1). Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
4. Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
5. Pregnant or breastfeeding females.
6. Major surgery within 4 weeks prior to C1D1.
7. Active, unstable cardiovascular function, as indicated by the presence of:

   1. Symptomatic ischemia, or
   2. Uncontrolled clinically significant conduction abnormalities (eg, patients with ventricular tachycardia on anti-arrhythmics are excluded; patients with first degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), or
   3. Congestive heart failure of New York Heart Association Class ≥3 or known left ventricular ejection fraction <40%, or
   4. Myocardial infarction within 3 months prior to C1D1.
8. Subjects with active hepatitis B virus (Hep B) are allowed if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 IU/ml prior to first dose of trial treatment. Subjects with untreated hepatitis C virus (HCV) are allowed.

   Subjects with Human Immunodeficiency Virus (HIV) who have CD4+ T-cell counts ≥ 350 cells/µL and no history of AIDS- defining opportunistic infections in the last year are allowed.
9. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment, including prior gastric bypass or bowel resection procedures.
10. Inability or unwillingness to take supportive medications such as anti-nausea and anti anorexia agents as recommended by the NCCN CPGO for antiemesis and anorexia/cachexia (palliative care).
11. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
12. Contraindication to any of the required concomitant drugs or supportive treatments.
13. Patients unwilling or unable to comply with the protocol, including providing 24-hour urine samples for urine protein electrophoresis at the required time points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-08-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate | Two years
  To evaluate the overall response rate achieved with physician's choice selinexor-based combination therapy as measured by International Myeloma Working Group criteria (based on Kumar et al 2016)

SECONDARY OUTCOMES:
MRD negative response rate | 2 years
  To evaluate the minimal residual disease negative response rate achieved with physician's choice selinexor-based combination therapy assessed via NGS or multiparametric flow cytometry with sensitivity of 10-5.
Progression Free Survival | 2 years
  To evaluate the duration of progression free survival achieved with physician's choice selinexor-based combination therapy
Overall Survival | 2 years
  To evaluate the duration of overall survival achieved with physician's choice selinexor-based combination therapy
Duration of Response | 2 years
  To evaluate the duration of response achieved with physician's choice selinexor-based combination therapy
Time to Next Treatment | 2 years
  To evaluate the time to next treatment achieved with physician's choice selinexor-based combination therapy
Safety and tolerability of selinexor | 2 years
  To evaluate safety and tolerability of selinexor in combination with partner backbone agents using occurrence, nature and severity of Adverse Events

OTHER OUTCOMES:
Reliability of My-DST testing to inform treatment choice | 2 years
  Rate of assay failure
Feasibility of My-DST testing to inform treatment choice | 2 years
  Rate of identification of preferred partner therapy or combination
Evaluation of My-DST related predictors of response | 2 years
  ORR in patients with concordance or discordance between My-DST results and physicians selected regimen

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sherbenou, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No